CLINICAL TRIAL: NCT06752824
Title: Evaluation of Analgesia Nociception Index Monitoring in Intracranial Surgery Anesthesia
Brief Title: Analgesia Nociception Index (ANI) in Intracranial Surgical Anesthesia
Acronym: ANI
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Neslihan Gunbay, RESEARCH ASSISTANT DOCTOR, Trakya University
Other Study IDs: TÜTF-BAEK 2020/406
Record Dates: First submitted 2024-12-20; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Pain, Postoperative; Analgesia; Supratentorial Brain Tumor; Infratentorial Neoplasms; Pituitary Neoplasms; Intraoperative Monitoring; Pain Monitoring
Keywords: INTRACRANIAL SURGERY; ENTROPY; ANI
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Infratentorial Neoplasms; Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- ANI GROUP: ANI MONITORING
  Interventions: Device: ANALGESIA NOCICEPTION INDEX MONITORING
- CONTROL GROUP: STANDARD MONITORING

INTERVENTIONS:
Device: ANALGESIA NOCICEPTION INDEX MONITORING — INTRACRANIAL SURGERY
  Other Names: ANI
  Groups: ANI GROUP

SUMMARY:
In our study, 75 patients aged 18-80 years, classified as ASA I-II risk groups, who underwent intracranial surgery performed by the Department of Neurosurgery at Trakya University Faculty of Medicine Hospital, were included. After the patients were positioned on the neurosurgical operating table, heart rate, systolic blood pressure, diastolic blood pressure, peripheral oxygen saturation, and entropy values were measured in all cases. Baseline values were recorded for patients who underwent ANI (Analgesia Nociception Index) monitoring. In both groups, entropy values were targeted to remain within the range of 40-60. In the ANI group, ANI values were maintained between 50-70.

Patients were divided into two groups based on the intraoperative monitoring method applied: the ANI group (n=38) and the control group (n=37). All patients underwent entropy monitoring, while ANI monitoring was exclusively used in the ANI group for pain management. In the ANI group, remifentanil infusion adjustments were made to keep ANI values within the 50-70 range.

This study aimed to compare perioperative opioid consumption, postoperative pain, and recovery from anesthesia in patients undergoing intracranial surgery who received general anesthesia and analgesia management guided by either entropy monitoring alone or a combination of entropy and ANI monitoring.

DETAILED DESCRIPTION:
In this study, we aimed to compare perioperative opioid consumption, postoperative pain, and recovery from anesthesia in patients undergoing intracranial surgery who were managed with general anesthesia and analgesia based on entropy monitoring or a combination of entropy and ANI monitoring during the intraoperative period.

A total of 75 patients aged between 18 and 80 years, classified as ASA I-II, who underwent intracranial surgery at Trakya University Medical Faculty Hospital between January 1, 2021, and January 1, 2024, were included in the study. Patients were divided into two groups based on the intraoperative monitoring techniques used: the ANI group (n=38) and the Control group (n=37). All patients underwent entropy monitoring during the operation. In the ANI group, ANI monitoring was additionally used for pain management.

The study recorded intraoperative data such as mean arterial pressure, heart rate, SpO2, end-tidal CO2, ANI, RE, SE values at baseline, induction, intubation, pin placement, skin incision, craniotomy, dura opening, bleeding control, pin removal, skin closure, and postoperatively. These values were measured at intervals of 5 minutes for the first 20 minutes, then every 10 minutes until 60 minutes, and every 30 minutes up to 180 minutes. Surgical type, anesthesia duration, the amount of erythrocyte suspension and fresh frozen plasma used based on intraoperative requirements, and anesthetic drugs (propofol, rocuronium, fentanyl) were recorded. The total remifentanil consumption was documented via the infusion pump.

Postoperative recovery in the recovery unit was evaluated using the Glasgow Coma Scale (GCS), the Ramsey Sedation Scale, and the duration with a Modified Aldrete Score (MAS) greater than 9. Pain was assessed using the Visual Analog Scale (VAS). VAS values were recorded at 1, 2, 4, 6, 12, and 24 hours. If VAS scores exceeded 4, intravenous paracetamol, tramadol, and meperidine were administered in stepwise treatment. The time to first analgesic use, postoperative analgesic consumption in the first 24 hours, and any postoperative complications were recorded.

Categorical variables were expressed as frequency distributions (number, percentage), and numerical variables were analyzed with descriptive statistics (mean, standard deviation). Differences between the two groups for categorical variables were examined using the independent samples t-test, Pearson correlation analysis was used to assess relationships between two numerical variables, and the Chi-square test was used to analyze relationships between two categorical variables. A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Patients between the ages of 18-80
* patients undergoing intracranial surgery

Exclusion Criteria:

* major comorbid diseases,
* patients using beta adrenergic blockers, clonidine,
* patients with pacemakers or significant arrhythmias (e.g. atrial fibrillation),
* patients using medications that affect sinus rhythm (atropine, ephedrine, glycopyrrolate),
* patients with chronic pain and cerebrovascular diseases,
* patients who will undergo planned postoperative ventilation,
* patients with chronic pain due to opioid medications, and patients with opioid addiction

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Seventy-five patients in ASA I-II risk group aged 18-80 who will undergo intracranial surgery by Brain and Nerve Surgery at Trakya University Faculty of Medicine Hospital will be included in the study.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
INTRAOPERATIVE OPIOID USE | during the surgery/procedure
  Lower dose opioid use during surgery is associated with more favorable outcomes in terms of postoperative pain and recovery scores.

CONTACTS AND LOCATIONS:
Overall Officials: SEVTAP HEKİMOĞLU ŞAHİN, Study Chair — Trakya University
Locations (1):
- Trakya Üniversitesi Tip Fakültesi, Edirne, Merkez, Turkey (Türkiye)